CLINICAL TRIAL: NCT06904040
Title: A Prospective, Single-Center, Single-Arm Clinical Study to Evaluate the Novel Humanized Cluster of Differentiation 38(CD38) Monoclonal Antibody (CM313) for the Treatment of Pemphigus
Brief Title: A Single-center Study of CM313 in Patients With Pemphigus
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Jianing Yang, Head of Dermatology, Sichuan Provincial People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CM313-IIS-PP01
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Pemphigus
MeSH Terms: conditions — Pemphigus | interventions — Glucocorticoids

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group 1 (Experimental)
  Interventions: Biological: CM313 injection; Biological: glucocorticoids

INTERVENTIONS:
Biological: CM313 injection — 600 mg (4 mL per vial), administer once at Week 0, 1, and 2, and then every 6 months thereafter or determined based on clinical assessment
Biological: glucocorticoids — Administer medium- or long-acting glucocorticoids 1-3 hours before injection

SUMMARY:
A prospective, single-center, single-arm clinical study aimed to explore the efficacy and safety of the anti-CD38 monoclonal antibody CM313 combined with low-dose glucocorticoids in patients with pemphigus.

ELIGIBILITY:
Inclusion Criteria:

* Clinical manifestations:① Flaccid blisters and bullae on the skin that are prone to rupture.② Persistent erosions formed after the rupture of blisters and bullae.③ Blisters or erosions on the mucous membranes.④ Positive Nikolsky's sign.
* Adult patients aged between 18 and 80 years old.
* Moderate - to - severe pemphigus vulgaris/foliaceus: According to the Pemphigus Disease Area Index (PDAI) score, a score of 9 - 24 indicates moderate severity, and a score of ≥25 indicates severe severity.

Exclusion Criteria:

* Pregnant or lactating women and women planning to conceive.
* Patients with known positive serology for HIV, syphilis, tuberculosis, hepatitis B, or hepatitis C in the active stage of the disease.
* Patients who have received intravenous cyclophosphamide injection, plasma exchange, or immunoadsorption therapy within 8 weeks before screening and enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-10-31 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy evaluation | up to 52 weeks
  The time to achieve disease control and consolidate the end

CONTACTS AND LOCATIONS:
Overall Officials: Jianing Yang, Principal Investigator — Sichuan Provincial People's Hospital
Locations (1):
- Sichuan Provincial People's Hospital, Chengdu, China